CLINICAL TRIAL: NCT03834961
Title: Larotrectinib (LOXO-101, NSC# 788607) for Previously Untreated TRK Fusion Pediatric Solid Tumors and TRK Fusion Relapsed Pediatric Acute Leukemias
Brief Title: Larotrectinib in Treating Patients With Previously Untreated TRK Fusion Solid Tumors and TRK Fusion Relapsed Acute Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1823; NCI-2019-00015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1823 (Other: Children's Oncology Group); ADVL1823 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-02-08 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Central Nervous System Neoplasm; Infantile Fibrosarcoma; Recurrent Acute Leukemia; Refractory Acute Leukemia; Solid Neoplasm
Keywords: Larotrectinib; TRK fusion; NTRK fusion; Infantile fibrosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — larotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (larotrectinib) (Experimental): Patients receive larotrectinib PO or by NG or G-tube BID on days 1-28. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity, or complete surgical resection of tumor.
  Interventions: Drug: Larotrectinib Sulfate

INTERVENTIONS:
Drug: Larotrectinib Sulfate — Given PO or via NG or G tube
  Other Names: ARRY 470 Sulfate; LOXO 101 Sulfate; LOXO-101 Sulfate; Vitrakvi

SUMMARY:
This phase II trial studies the side effects and how well larotrectinib works in treating patients with previously untreated TRK fusion solid tumors and TRK fusion acute leukemia that has come back. Larotrectinib may stop the growth of cancer cells with TRK fusions by blocking the TRK enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR) of children with infantile fibrosarcoma (IFS) treated with neoadjuvant larotrectinib prior to local control.

SECONDARY OBJECTIVES:

I. To determine event-free survival (EFS), overall survival (OS), and duration of response (DoR) of children with IFS treated with neoadjuvant larotrectinib prior to local control.

II. To determine the ORR, EFS, OS, and DoR of children with newly diagnosed TRK fusion solid tumors other than IFS treated with neoadjuvant larotrectinib prior to local control.

III. To describe the toxicity of larotrectinib in children with solid tumors and acute leukemia.

IV. To determine the percentage of patients with TRK fusion solid tumors with detectable circulating tumor deoxyribonucleic acid (DNA) at baseline and after 2 weeks, 4 weeks, 24 weeks of treatment, at the time of discontinuation of larotrectinib therapy, and at progression.

EXPLORATORY OBJECTIVES:

I. To determine the EFS, OS, and DoR of children with TRK fusion solid tumors other than IFS treated with adjuvant larotrectinib following upfront surgery with positive margins after neoadjuvant larotrectinib.

II. To determine the EFS, OS, and DoR of children with TRK fusion solid tumors who experience a complete response to larotrectinib and subsequently discontinue larotrectinib therapy.

III. To determine the remission induction rate for patients with recurrent/refractory TRK fusion leukemia when treated with larotrectinib.

IV. To evaluate the surgical morbidity and extent of resection of initially unresectable tumors in patients with TRK fusion solid tumors who undergo surgical resection following neoadjuvant larotrectinib.

V. To evaluate mechanisms of response and resistance to larotrectinib in children with TRK fusion cancers.

VI. To evaluate the morphologic features of TRK fusion solid tumors at time of initial biopsy to further define criteria for pathologic diagnosis of these tumors.

VII. To evaluate immunohistochemistry for pan-TRK as a screening method for TRK fusion tumors and in resection specimens following neoadjuvant treatment with larotrectinib.

VIII. To evaluate the histologic response to larotrectinib in resection specimens following neoadjuvant treatment.

IX. To evaluate circulating tumor DNA for the detection of the emergence of resistance mutations and recurrence in patients with TRK fusion solid tumors treated with larotrectinib.

X. To evaluate the ratio of cerebrospinal fluid (CSF) to concurrent plasma concentrations of larotrectinib in patients with leukemia.

XI. To evaluate the change in neurocognitive/behavioral functioning over time between baseline and 5 years post-diagnosis of patients treated on this protocol using parent-reported adaptive functioning (Adaptive Behavior Assessment System [ABAS]-III General Adaptive Composite), executive function (Behavior Rating Inventory of Executive Function Scales-Preschool Version [BRIEF-P] or BRIEF-2 Global Executive Composite Score), psychosocial functioning (Behavior Assessment System for Children [BASC]-3 Internalizing, Externalizing and Behavioral Symptoms Indices) and quality of life (Pediatric Quality of Life Inventory [PedsQL] Total score).

OUTLINE:

Patients receive larotrectinib orally (PO) or by nasogastric (NG) or gastric tube (G-tube) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity. Patients whose tumors shrink sufficiently while taking larotrectinib may undergo surgical resection of their tumor while on study.

After completion of study treatment, patients are followed up at 3, 6, 12, 18, 24, 30, 36, and 48 months and annually thereafter for up to 5 years from the date of study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be =< 30 years of age at the time of study entry
* COHORT A: Patients must have a histologic diagnosis of infantile fibrosarcoma with an NTRK1, NTRK2, or NTRK3 fusion identified in a Clinical Laboratory Improvement Act/College of American Pathologists (CLIA/CAP) certified laboratory. Fusions may be identified by fluorescence in situ hybridization (FISH) or molecular techniques (reverse transcriptase-polymerase chain reaction [RT-PCR] using primers flanking the fusion junction or next generation sequencing). For fusions identified by FISH, an ETV6 rearrangement is sufficient for eligibility in Cohort A. Identification of the upstream TRK fusion partner is not required.
* COHORT B: Patients must have a histologic diagnosis of any solid tumor other than infantile fibrosarcoma, including central nervous system (CNS) tumors but excluding high grade gliomas. An NTRK1, NTRK2, or NTRK3 fusion must be identified in a CLIA/CAP certified laboratory. Fusions may be identified by FISH or molecular techniques (RT-PCR using primers flanking the fusion junction or next generation sequencing). For fusions identified by FISH, there must be an identified rearrangement in NTRK1, NTRK2, or NTRK3 (e.g., an ETV6 rearrangement is not sufficient for eligibility) unless the patient has a diagnosis of congenital mesoblastic nephroma in which case an ETV6 rearrangement is sufficient for eligibility. Identification of the upstream TRK fusion partner is not required.
* COHORT C: Patients must have a histologic diagnosis of relapsed or refractory acute leukemia with an NTRK1, NTRK2, or NTRK3 fusion identified in a CLIA/CAP certified laboratory. Fusions may be identified by FISH or molecular techniques (RT-PCR using primers flanking the fusion junction or next generation sequencing). For fusions identified by FISH, there must be an identified rearrangement in NTRK1, NTRK2, or NTRK3 (e.g., an ETV6 rearrangement is not sufficient for eligibility). Identification of the upstream TRK fusion partner is not required.
* SOLID TUMORS (COHORTS A AND B): Patients must have measurable disease. Patients must have disease that cannot be completely resected without a predicted functional, neurologic, or significant cosmetic deficit in the opinion of the investigator.
* LEUKEMIA (COHORT C): Patients must have >= 5% blasts in the bone marrow. Extramedullary disease is permitted.
* Patients must have a Lansky or Karnofsky performance status score of >= 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age. NOTE: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* COHORTS A AND B: No prior anti-cancer therapy, including radiotherapy, other than surgical resection is permitted.

  * Patients who experience recurrence after surgery alone and no other anti-cancer therapy will be eligible.
  * If not eligible due to prior anticancer therapy, patients may be eligible for the larotrectinib arm of Pediatric MATCH (APEC1621A) or treatment with commercial larotrectinib off study.
* COHORT C: Patients with relapsed leukemia (Cohort C) must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately.

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive.

    * A waiting period prior to enrollment is not required for patients receiving standard cytotoxic maintenance chemotherapy (i.e., corticosteroid, vincristine, thioguanine [6MP], and/or methotrexate).
    * A waiting period is not required for patients receiving a single dose of intrathecal methotrexate, hydrocortisone, and/or cytarabine within 7 days prior to enrollment.
    * >= 14 days must have elapsed after the completion of other cytotoxic therapy, with the exception of hydroxyurea, for patients not receiving standard maintenance therapy. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy.

      * Note: Cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy.
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil [ANC] counts): >= 7 days after the last dose of agent.
  * Anti-cancer agents that are antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1. There is an exception for blinatumomab infusions, for which patients must have been off for at least 3 days and all drug related toxicity must have resolved to grade 2 or lower as outlined in the inclusion/exclusion criteria.
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid. A waiting period prior to enrollment is not required for patients receiving corticosteroid for leukemia therapy/cytoreduction.
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator.
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors ).
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD).
    * Autologous stem cell infusion including boost infusion: >= 42 days.
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial BM radiation.
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody): >= 42 days after systemically administered radiopharmaceutical therapy.
  * Patients must not have received prior exposure to TRK inhibitors (including larotrectinib, LOXO-195, entrectinib, lorlatinib, crizotinib, or lestaurtinib).
* For patients with solid tumors without known bone marrow involvement: Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days prior to enrollment).
* For patients with solid tumors without known bone marrow involvement: Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* For patients with solid tumors without known bone marrow involvement: Hemoglobin >= 8.0 g/dL at baseline (within 7 days prior to enrollment) (may receive red blood cell [RBC] transfusions).
* Patients with solid tumors with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts above (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity.
* For patients with leukemia: Platelet count >= 20,000/mm^3 (within 7 days prior to enrollment) (may receive platelet transfusions; must not be known to be refractory to red cell or platelet transfusion).
* For patients with leukemia: Hemoglobin >= 8.0 g/dL at baseline (within 7 days prior to enrollment) (may receive RBC transfusions; must not be known to be refractory to red cell or platelet transfusion).
* For patients with leukemia: These patients must not be known to be refractory to red cell or platelet transfusion.
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * 1 month to < 6 months (male 0.4 mg/dL, female 0.4 mg/dL)
  * 6 months to < 1 year (male 0.5 mg/dL, female 0.5 mg/dL)
  * 1 to < 2 years (male 0.6 mg/dL, female 0.6 mg/dL)
  * 2 to < 6 years (male 0.8 mg/dL, female 0.8 mg/dL)
  * 6 to < 10 years (male 1 mg/dL, female 1 mg/dL)
  * 10 to < 13 years (male 1.2 mg/dL, female 1.2 mg/dL)
  * 13 to < 16 years (male 1.5 mg/dL, female 1.4 mg/dL)
  * >= 16 years (male 1.7 mg/dL, female 1.4 mg/dL)

    * For patients < 1 month of age, serum creatinine levels must be < 1.5 x the treating institution's creatinine upper limit of normal (ULN) for patients < 1 month of age or the creatinine clearance or radioisotope GFR must be >= 70 mL/min/1.73 m^2.
* Patients with solid tumors: Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment). After approval of the study chair or designee, infants with a higher total bilirubin due to physiologic or breast milk jaundice are eligible if the conjugated (direct) bilirubin is =< 2 mg/dL.
* Patients with solid tumors: Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment). For the purpose of this study, the ULN for SGPT is 45 U/L.
* Patients with solid tumors: Serum albumin >= 2 g/dL (within 7 days prior to enrollment).
* Patients with leukemias: Conjugated (direct) bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment).
* Patients with leukemias: SGPT (ALT) =< 225 U/L (within 7 days prior to enrollment). For the purpose of this study, the ULN for SGPT is 45 U/L.
* Patients with leukemias: Serum albumin >= 2 g/dL (within 7 days prior to enrollment).
* Patients with seizure disorder may be enrolled if on a stable antiepileptic regimen for >= 14 days and well controlled.
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5) except tendon reflex decreased resulting from prior therapy must be =< grade 2.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Female patients of reproductive potential may not participate unless they have agreed to use a highly effective contraceptive method for the duration of study therapy and for at least one month after the final dose of larotrectinib. Males of reproductive potential with a non-pregnant female partner of child-bearing potential must use a highly effective contraception for the duration of the study and for at least one month after the final dose of larotrectinib. Because of the unknown risk of larotrectinib in nursing infants, nursing women should discontinue breastfeeding during treatment with larotrectinib and for 3 days following the final dose.
* Patients with solid tumors, including CNS tumors, requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. Patients with leukemia may receive systemic corticosteroids for cytoreduction up to 24 hours prior to the start of protocol therapy. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid.
* Patients who are currently receiving another investigational drug are not eligible.
* Patients who are currently receiving other anti-cancer agents are not eligible [except leukemia patients receiving corticosteroids or hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy]. Patients with leukemia should receive a single dose of intrathecal cytarabine, hydrocortisone, and/or methotrexate within 7 days prior to Day 1 of Cycle 1 at the time of the baseline lumbar puncture.
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial.
* Patients currently receiving a strong CYP3A4 inducer or inhibitor are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study. Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed.
* Patients with malabsorption syndrome or other conditions that significantly limit enteral absorption are not eligible.
* Patients who are unable to swallow capsules or liquid and do not have gastric access via a nasogastric or gastrostomy tube are not eligible.
* Patients who have an uncontrolled infection are not eligible.
* Patients who have received prior solid organ transplantation are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
* Patients with high grade gliomas (HGG) are not eligible.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2027-07-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore W Laetsch, Principal Investigator — Children's Oncology Group
Locations (80):
- United States (78):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - IWK Health Centre, Halifax, Nova Scotia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Laetsch TW, Voss S, Ludwig K, Hall D, Barkauskas DA, DuBois SG, Ronan J, Rudzinski ER, Memken A, Robinson K, Sorger J, Reid JM, Bhatla T, Crompton BD, Church AJ, Fox E, Weigel BJ. Larotrectinib for Newly Diagnosed Infantile Fibrosarcoma and Other Pediatric NTRK Fusion-Positive Solid Tumors (Children's Oncology Group ADVL1823). J Clin Oncol. 2025 Apr;43(10):1188-1197. doi: 10.1200/JCO-24-01854. Epub 2024 Dec 9. PMID 39652801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Zero patients were assigned to Cohort C
Groups:
- Cohort A: Patients with infantile fibrosarcoma with an NTRK1, NTRK2, or NTRK3 fusion identified
- Cohort B: Patients with solid tumors including CNS tumors, with an NTRK1, NTRK2, or NTRK3 fusion identified
- Cohort C: Patients with a histologic diagnosis of relapsed or refractory acute leukemia with an NTRK1, NTRK2, or NTRK3 fusion identified
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 18 | 15 | 0
Completed | 17 | 13 | 0
Not Completed | 1 | 2 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Zero patients were assigned to Cohort C
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 18 | 15 | 0 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 14 |  | 32
  Between 18 and 65 years | 0 | 1 |  | 1
  >=65 years | 0 | 0 |  | 0
Age, Continuous [Median (Full Range); unit: years] | 0.2 [0.0 to 4.6] | 9.4 [0.4 to 20.9] |  | 0.7 [0.0 to 20.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 |  | 14
  Male | 12 | 7 |  | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 |  | 5
  Not Hispanic or Latino | 10 | 12 |  | 22
  Unknown or Not Reported | 4 | 2 |  | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 2 | 3 |  | 5
  White | 13 | 10 |  | 23
  More than one race | 2 | 0 |  | 2
  Unknown or Not Reported | 1 | 2 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Children With Infantile Fibrosarcoma (IFS) Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: A responder is defined as a patient who achieves a best response of partial response (PR) or complete response (CR) on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed accounting for the two-stage design.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A
Number analyzed (Participants) | 18
percentage of patients | 94.4 [80.1 to 97.0]

2. Secondary Outcome: Event-free Survival (EFS) of Children With IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: The Kaplan-Meier method will be used to estimate 1-year EFS, defined as the time from study entry until last contact, relapse, secondary malignancy, or death.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A
Number analyzed (Participants) | 18
percentage of patients | 94.4 [66.6 to 99.2]

3. Secondary Outcome: Overall Survival (OS) of Children With IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: The Kaplan-Meier method will be used to estimate 1-year OS, defined as the time from study entry until last contact or death.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A
Number analyzed (Participants) | 18
percentage of patients | 100 [100.0 to 100.0]

4. Secondary Outcome: Duration of Response (DoR) of Children With IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: Will be defined among patients with a confirmed best response of either PR and CR. Will be computed as the time from first observation of either PR or CR until either the first observation of progressive disease (PD) (event) or last known observation of the patient (censored observation).
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: years
Groups:
- Cohort A: Patients with infantile fibrosarcoma with an NTRK1, NTRK2, or NTRK3 fusion identified with overall best response of Complete Response or Partial Response.
Arm/Group | Cohort A
Number analyzed (Participants) | 17
years | 2.1 [0.4 to 4.2]

5. Secondary Outcome: ORR of Children and Adults With Newly Diagnosed TRK Fusion Solid Tumors Other Than IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: A responder is defined as a patient who achieves a best response of PR or CR on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed accounting for the two-stage design.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort B
Number analyzed (Participants) | 15
percentage of patients | 60 [32.3 to 83.7]

6. Secondary Outcome: EFS of Children and Adults With Newly Diagnosed TRK Fusion Solid Tumors Other Than IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: as for outcome 2
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B
Number analyzed (Participants) | 15
percentage of participants | 93.3 [61.3 to 99.0]

7. Secondary Outcome: OS of Children and Adults With Newly Diagnosed TRK Fusion Solid Tumors Other Than IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: as for outcome 3
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort B
Number analyzed (Participants) | 15
percentage of patients | 93.3 [61.3 to 99.0]

8. Secondary Outcome: DoR of Children With Newly Diagnosed TRK Fusion Solid Tumors Other Than IFS Treated With Neoadjuvant Larotrectinib Prior to Local Control
Description: Will be defined among patients with a confirmed best response of either PR and CR. Will be computed as the time from first observation of either PR or CR until either the first observation of PD (event) or last known observation of the patient (censored observation).
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: years
Groups:
- Cohort B: Patients with solid tumors, including CNS tumors, with an NTRK1, NTRK2, or NTRK3 fusion identified with overall best response of Complete Response or Partial Response.
Arm/Group | Cohort B
Number analyzed (Participants) | 9
years | 2.9 [0.2 to 4.8]

9. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Will report the percentage of patients within each disease stratum who experienced a grade 3 or higher toxicity with attribution of possible, probable, or definite while on protocol therapy or within 30 days of the last dose of therapy. Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Through 30 days after treatment, a mean of 12.6 months
Population: Zero patients were assigned to Cohort C
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 18 | 15 | 0
percentage of patients | 44.4 [21.5 to 69.2] | 20 [4.3 to 48.1] |

10. Secondary Outcome: Percentage of Patients With TRK Fusion Solid Tumors With Detectable Circulating Tumor Deoxyribonucleic Acid (ctDNA)
Description: The percentage of ctDNA and frequency with which patients have detectable ctDNA prior to the start of therapy and at times during therapy when subsequent serial samples are obtained (2 weeks, 4 weeks, 24 weeks of treatment, at the time of discontinuation of larotrectinib therapy, and at progression) will be calculated.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: Through 30 days after treatment, a mean of 12.6 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 1/18 | 1/15 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/18 | 1/15 | 0/0
Other Adverse Events (participants affected / at risk) | 9/18 | 5/15 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=18) | Cohort B (N=15) | Cohort C (N=0)
Optic nerve disorder (Eye disorders) | 0 | 1 | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | NA
Sepsis (Infections and infestations) | 1 | 0 | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | NA
Irritability (Psychiatric disorders) | 1 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=18) | Cohort B (N=15) | Cohort C (N=0)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | NA
Sinus tachycardia (Cardiac disorders) | 0 | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | NA
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | NA
Alanine aminotransferase increased (Investigations) | 0 | 2 | NA
Aspartate aminotransferase increased (Investigations) | 0 | 2 | NA
Blood bilirubin increased (Investigations) | 1 | 0 | NA
Lymphocyte count decreased (Investigations) | 0 | 1 | NA
Neutrophil count decreased (Investigations) | 5 | 2 | NA
Weight gain (Investigations) | 0 | 2 | NA
Weight loss (Investigations) | 1 | 0 | NA
White blood cell decreased (Investigations) | 0 | 2 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | NA
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | NA
Insomnia (Psychiatric disorders) | 0 | 1 | NA
Hypertension (Vascular disorders) | 2 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT03834961/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT03834961/ICF_000.pdf